CLINICAL TRIAL: NCT04277676
Title: Reliability and Validity of Turkish Version of Knee Injury and Osteoarthritis Outcome Score-12
Acronym: KOOS-12
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Leyla Ataş Balcı, Assist. Prof, Bahçeşehir University
Other Study IDs: 22481095-020-4023
Record Dates: First submitted 2020-02-06; First posted 2020-02-20 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Osteo Arthritis Knee
Keywords: KOOS; Knee; Osteoarthritis; Patient-reported outcome measures; Psychometrics
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Approximately 120 patients who have been diagnosed with knee osteoarthritis but have not previously operated due to this disease and who are in Kellgren Lawrence stage 2 and 3 will be compared with the KOOS scale and Short Form-36 (Short Form-36: SF-36) scales to investigate the validity and reliability of the Turkish version of KOOS-12.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic degenerative disease characterized by the loss of articular cartilage, causing destruction in periarticular bone tissue, leading to a decrease in daily life and quality of life due to pain despite its slow progression.

When the knee osteoarthritis Looking at the prevalence among people living in Turkey, compared to males more can be seen, 14.8% of the 50 and older population in knee OA incidence, 22.5% of the incidence in women, while men were determined to be 8%.

Risk factors that affect the development of knee OA include obesity, traumas, chondrocalcinosis, nutritional factors, genetics, smoking, estrogen replacement, muscular weakness, and professional or sports activities. The individual with knee OA especially; It is applied to the physician with the complaints of increased pain during walking, climbing and climbing stairs, stiffness in the joint, crepitation and limited range of motion.

Diagnosis is determined based on knee OA, clinical and radiological evaluations; According to the radiological changes seen, the stage of the disease is determined by Kellgren Lawrence staging (Stage 0-4). Purposes in the treatment of knee OA; patient education, pain control, increasing functionality and reducing the impact of disability on daily life. The optimal treatment approach involves the application of non-pharmacological and pharmacological treatments together.

Functional evaluation methods are of great importance in planning the right treatment approach and evaluating treatment effectiveness due to the negative impact of individuals on daily life activities. Functional evaluation of the individual; daily life activities, professional activities, leisure activities, social relationships and their skills in performing these tasks are carried out with objective, generic or disease-specific scales. Various scales have been developed in individuals with knee OA that allow an objective evaluation of functions. Among these scales, Western Ontario and McMaster Universities Osteoarthritis Index (Western Ontario and McMaster Universities Osteoarthritis Index: WOMAC), Lequesne Index, Knee-Hip Osteoarthritis Life Quality Scale (Osteoarthritis of Knee Hip Quality Of Life Questionnaire: OAKHQOL), Knee osteoarthritis and Knee Injury and Knee Injury and Osteoarthritis Outcome Score: KOOS.

These questionnaires, which are reported by the patients, are not routinely used in the clinic due to the length of the questionnaires, which are used to determine the problems caused by joint problems in daily life and quality of life. Therefore, patient-based scales that can be used in the clinic should be short, and include questions that can evaluate pain, function and quality of life. Although the short form of the KOOS questionnaire has been developed, KOOS-PS only measures the effects of knee osteoarthritis on physical function. Consisting of 12 questions considering that the KOOS scale is long in routine, clinic use; A short form of KOOS-12 was created, which included the assessment sections of pain, function and knee-specific quality of life. The application of the KOOS-12 scale takes 2 minutes. The short form of KOOS-12 was found to be a valid and reliable scale in individuals who underwent total knee arthroplasty. The purpose of our study; Turkish reliability and validity of the Knee Osteoarthritis and Knee Injury and Osteoarthritis Result Score-12 scale.

ELIGIBILITY:
Inclusion Criteria:

* The study resides in the province of Istanbul
* 18 years and older
* Who have been diagnosed with knee osteoarthritis
* In Kellgren Lawrence Staging; Stage 2 and 3 detected
* Not operated after knee osteoarthritis after diagnosis
* Literate
* 120 individuals who agree to participate in the study will be included. For the validity of the questionnaire, it must be applied to at least 10 times the number of questions in the questionnaire. In this context, it is planned to be included in the study with at least 120 people.

Exclusion Criteria:

* Those diagnosed with hip and ankle OA
* Those with neurological diseases affecting their lower extremities
* Those with knee pain due to rheumatoid arthritis, anterior cruciate ligament injury and menisectomy
* Those who had a total knee arthroplasty operation in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In determining the individuals who will participate in the study; face to face interviews and social media groups (whatsapp, facebook, instagram etc.) will be used. Individuals diagnosed with osteoarthritis by the physician at the Alptekin Physical Therapy Clinic will be included.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score-12 (KOOS-12) | change from baseline activities od daşly living at 2 weeks
  Scale; It consists of three parts: pain (4 items), function (4 items) and knee-specific quality of life (4 items). KOOS-12; in pain sub-item; In the sub-item of walking on a flat ground, going up and down stairs, sitting-reaching, function and daily life; There are patient-specific questions in the sub-item of quality of life, sitting up, standing, getting in and out of the car, turning the affected knee. The total scores obtained from the items in the KOOS-12 scale are calculated and the average of the total score is taken from the three sub-dimensions. If any of the three sub-item scores are missing, the average score cannot be calculated.
Knee injury and Osteoarthritis Outcome Score (KOOS) | change from baseline activities od daşly living at 2 weeks
  It is a questionnaire designed by Roos et al. From the Likert 3.0 version of the WOMAC osteoarthritis index to evaluate the pain, functional status, daily life activity and quality of life of patients with knee osteoarthritis (Roos EM. et al. 1998). Scale; consists of five subgroups and 42 questions: pain, string-related quality of life, daily life activities, sports and leisure activities. Individuals score the questions between 0-4 according to the 5-point Likert scale, based on the symptoms felt in the knee, taking into account the past week. While 100 points indicate that there are no symptoms in the scale, 0 points indicate that there are severe symptoms. The subscale score is calculated by dividing the average scores of each sub-dimension separately into 4. The Turkish validity and reliability study of the scale was conducted. (Sabırlı F. et al. 2007). It takes 10 minutes to apply the scale (Roos EM. et al. 2003, Paker N. et al. 2007).
Short Form-36 (SF-36) | change from baseline activities od daşly living at 2 weeks
  It is a scale that is used to evaluate the overall quality of life consisting of eight sub-scales and 36 questions and allows the individual to evaluate himself. Scale; physical function, physical role, emotional role, pain, vitality, general health and mental health sub-dimensions. Each subscale is scored between 0-100 and "0" indicates the lowest and "100" shows the best quality of life. The questionnaire has Turkish validity and reliability (Kocyigit H. et al. 1999).

CONTACTS AND LOCATIONS:
Locations (1):
- Alptekin Physical Therapy and Rehabilitation Clinic, Istanbul, Beşiktaş/İstanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Result] Felson DT. The epidemiology of knee osteoarthritis: results from the Framingham Osteoarthritis Study. Semin Arthritis Rheum. 1990 Dec;20(3 Suppl 1):42-50. doi: 10.1016/0049-0172(90)90046-i. PMID 2287948
- [Result] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Result] Scott DL, Garrood T. Quality of life measures: use and abuse. Baillieres Best Pract Res Clin Rheumatol. 2000 Dec;14(4):663-87. doi: 10.1053/berh.2000.0106. PMID 11092795
- [Result] Recommendations for the medical management of osteoarthritis of the hip and knee: 2000 update. American College of Rheumatology Subcommittee on Osteoarthritis Guidelines. Arthritis Rheum. 2000 Sep;43(9):1905-15. doi: 10.1002/1529-0131(200009)43:93.0.CO;2-P. No abstract available. PMID 11014340
- [Result] Bellamy N. WOMAC: a 20-year experiential review of a patient-centered self-reported health status questionnaire. J Rheumatol. 2002 Dec;29(12):2473-6. No abstract available. PMID 12465137
- [Result] Faucher M, Poiraudeau S, Lefevre-Colau MM, Rannou F, Fermanian J, Revel M. Assessment of the test-retest reliability and construct validity of a modified Lequesne index in knee osteoarthritis. Joint Bone Spine. 2003 Dec;70(6):521-5. doi: 10.1016/s1297-319x(03)00070-8. PMID 14667565
- [Result] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Result] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Rheum Dis Clin North Am. 2008 Aug;34(3):515-29. doi: 10.1016/j.rdc.2008.05.007. PMID 18687270
- [Result] Hunter DJ, Lo GH. The management of osteoarthritis: an overview and call to appropriate conservative treatment. Rheum Dis Clin North Am. 2008 Aug;34(3):689-712. doi: 10.1016/j.rdc.2008.05.008. PMID 18687278
- [Result] Gandek B, Roos EM, Franklin PD, Ware JE Jr. A 12-item short form of the Knee injury and Osteoarthritis Outcome Score (KOOS-12): tests of reliability, validity and responsiveness. Osteoarthritis Cartilage. 2019 May;27(5):762-770. doi: 10.1016/j.joca.2019.01.011. Epub 2019 Feb 1. PMID 30716536
- See also: Şencan H. Sosyal ve davranışsal ölçümlerde güvenilirlik ve geçerlilik. 1.Baskı. Ankara: Seçkin Yayınevi, 2005; 384-386 — https://www.ders.es/guvenilirlik_gecerlilik.pdf
- See also: Granger CV, Black T, Braun SL. Quality and outcome measures for medical rehabilitation. In: Braddom RL (Ed). Physical Medicine and Rehabilitation. 3rd Edition. China, Saunders Elseiver, China, 2007, pp 151-64. — http://static.ato.org.tr/fs/4f4f77c367cde9271f000002/hekimler_icin_temel_geriatri_kitabi.pdf
- See also: Kutsal Y, Kara M. Diz Osteoartriti. M S, editor. İstanbul: Nobel Tıp Kitabevi; 2007. s. 149-161. — https://dergipark.org.tr/tr/pub/hunhemsire/issue/44118/544133
- See also: Guler Uysal F, Başaran S. Knee oteoarthritis Turl J Phys Med Rehab.2009;55 Suppl 1;1-7 — http://www.ftrdergisi.com/abstract.php?lang=tr&id=3086
- See also: Karakoç FY, Dönmez L. Ölçek Geli̇şti̇rme Çalışmalarında Temel İlkeler. Tıp Eğitimi Dünyası. 2014; 40: 39-49 — http://dergipark.org.tr/en/download/article-file/199275
- See also: The European Musculoskeletal Conditions Surveillance. Musculoskeletal health in europe report v5.0 (online) 2016: (3 screens). Available from: URL: http://www.eumusc.net/myUploadData/files/Musculoskeletal%20Health%20in%20 Europe%20Report%20v5.pdf. — http://dergipark.org.tr/tr/pub/hunhemsire/article/544133
- See also: Göksoy T, Romatizmal Hastalıkların Tanı ve Tedavisi. İç: Cerrahoğlu L, Kokino S, editör. Osteoartrit. Yüce Yay; 2002. S.379- 405 — https://www.journalagent.com/kafkas/pdfs/KJMS_8_50_133_142.pdf
- See also: Kocyigit H, Aydemir O, Fisek G, et al. Validity and reliability of Turkish version of SF-36. İlaç ve Tedavi Dergisi. 1999;12:102-106. — http://jsurgmed.com/tr/download/article-file/419612